CLINICAL TRIAL: NCT05116514
Title: Evaluation of the Impact of Case Manager Intervention on the 3-year Psychotic Episode Recurrence Rate in Patients Aged 16 to 30 Years With a First Psychotic Episode. Randomized, Open-label, Multicenter Controlled Study With Blinded Evaluation.
Brief Title: Evaluation of the Impact of Case Manager Intervention on the 3-year Psychotic Episode Recurrence Rate in Patients Aged 16 to 30 Years With a First Psychotic Episode.
Acronym: PEPsy-CM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PREPS/2018/AS-01
Record Dates: First submitted 2021-10-05; First posted 2021-11-11 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Psychotic Episode
MeSH Terms: interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case manager group (Experimental)
  Interventions: Other: Case management
- Control (No Intervention)

INTERVENTIONS:
Other: Case management — Regular and personalized follow-up by a case manager using a "case management" approach, updated every 3 months
  Arms: Case manager group

SUMMARY:
The study investigators hypothesize that the intervention of case managers specifically trained in case management of early psychosis will change the paradigm of care of a first psychotic episode from the current organization of the care system. Indeed, the creation of specific services for emerging psychotic disorders cannot easily be generalized throughout the country and requires specific funding. The intervention of case managers according to the recommendations of good practices will make it possible to propose the fundamental principles of early intervention to young patients and their families on a large scale throughout the territory, namely: personalized and proactive accompaniment, psycho-education of the pathology and treatments, involvement and support of the families, and support for socio-professional reintegration

ELIGIBILITY:
Inclusion Criteria:

* The patient or their close relative must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is available for a 3-year follow-up.
* Patient is managed in a psychiatric service (consultation or hospitalization) for a first episode psychosis defined by:

  * Presence of positive psychotic symptoms (delusion(s) and/or hallucination(s) and/or conceptual disorganization) evolving for at least one week, either daily or at least 3 times per week for at least one hour per occasion ;
  * Never having taken a neuroleptic treatment with antipsychotic aim (except for an antipsychotic treatment started for the current episode for example by the general practitioner before being referred to psychiatry);
  * A disorder meeting the DSM 5 criteria from the following list: delusional disorder, brief psychotic disorder greater than 7 days, schizophreniform disorder, schizophrenia, schizoaffective disorder, substance-induced psychotic disorder greater than 7 days, other specific or nonspecific schizophrenic spectrum disorder or other psychotic disorder, bipolar I or II disorder with congruent and non-mood congruent psychotic features, bipolar disorder with congruent and non-mood congruent psychotic features induced by a substance, major depressive disorder with congruent and non-mood congruent psychotic features.
* Inclusion should be within the first 3 months of care for first episode psychosis in the psychiatric service.
* At the time of inclusion, the psychotic symptomatology observed during the first episode psychosis may still be present or in remission.

Exclusion Criteria:

* The subject is participating in another category I interventional study, or is in a period of exclusion determined by a previous study
* The subject, or one of the parents for minor patients, refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patients has an IQ less than or equal to 55
* The patient has a first psychotic episode linked to a psychotic problem triggered by a medication of other medical condition
* The patient is pregnant or breastfeeding

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 256 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with recurrence of psychotic episode at least once between groups | 3 years
  Recurrence of the psychotic episode will be defined as psychiatric hospitalization with a diagnosis of psychotic disorder and/or the presence of positive psychotic symptoms according to the Positive and Negative Symptom Scale (PANSS) ≥ 4 for item P1 (delusions) and/or P2 (conceptual disorganization) and/or P3 (hallucination)) over a period of at least one week.

SECONDARY OUTCOMES:
Evaluate the impact of the intervention on the number of recurrences of psychiatric hospitalization per patient | 1 year
  number
Evaluate the impact of the intervention on the number of recurrences of psychiatric hospitalization per patient | 2 years
  number
Evaluate the impact of the intervention on the number of recurrences of psychiatric hospitalization per patient | 3 years
  number
Evaluate the impact of the intervention on the number of psychiatric hospitalizations per patient | 1 year
  number
Evaluate the impact of the intervention on the number of psychiatric hospitalizations per patient | 2 years
  number
Evaluate the impact of the intervention on the number of psychiatric hospitalizations per patient | 3 years
  number
Evaluate the impact of the intervention on the duration of psychiatric hospitalization per patient | 1 year
  days/weeks/months
Evaluate the impact of the intervention on the duration of psychiatric hospitalization per patient | 2 years
  days/weeks/months
Evaluate the impact of the intervention on the duration of psychiatric hospitalization per patient | 3 years
  days/weeks/months
Percentage per patient of medical and caregiving appointments honored between groups | Inclusion
  %
Percentage per patient of medical and caregiving appointments honored between groups | 6 months
  %
Percentage per patient of medical and caregiving appointments honored between groups | 1 year
  %
Percentage per patient of medical and caregiving appointments honored between groups | 18 months
  %
Percentage per patient of medical and caregiving appointments honored between groups | 2 years
  %
Percentage per patient of medical and caregiving appointments honored between groups | 2.5 years
  %
Percentage per patient of medical and caregiving appointments honored between groups | 3 years
  %
Type of hospital admission (voluntary versus involuntary) between groups | Inclusion
  % voluntary versus involuntary
Type of hospital admission (voluntary versus involuntary) between groups | 6 months
  % voluntary versus involuntary
Type of hospital admission (voluntary versus involuntary) between groups | 1 year
  % voluntary versus involuntary
Type of hospital admission (voluntary versus involuntary) between groups | 18 months
  % voluntary versus involuntary
Type of hospital admission (voluntary versus involuntary) between groups | 2 years
  % voluntary versus involuntary
Type of hospital admission (voluntary versus involuntary) between groups | 2.5 years
  % voluntary versus involuntary
Type of hospital admission (voluntary versus involuntary) between groups | 3 years
  % voluntary versus involuntary
Unscheduled discharge from care between groups | Inclusion
  Defined by a break in follow-up organized by the referring care team for more than 30 days
Unscheduled discharge from care between groups | 6 months
  Defined by a break in follow-up organized by the referring care team for more than 30 days
Unscheduled discharge from care between groups | 1 year
  Defined by a break in follow-up organized by the referring care team for more than 30 days
Unscheduled discharge from care between groups | 18 months
  Defined by a break in follow-up organized by the referring care team for more than 30 days
Unscheduled discharge from care between groups | 2 years
  Defined by a break in follow-up organized by the referring care team for more than 30 days
Unscheduled discharge from care between groups | 2.5 years
  Defined by a break in follow-up organized by the referring care team for more than 30 days
Unscheduled discharge from care between groups | 3 years
  Defined by a break in follow-up organized by the referring care team for more than 30 days
Treatment compliance between groups | Inclusion
  item 13 of the Health of the Nation Outcome Scales (HoNOS, hetero-assessment)
Treatment compliance between groups | 6 months
  item 13 of the Health of the Nation Outcome Scales (HoNOS, hetero-assessment)
Treatment compliance between groups | 1 year
  item 13 of the Health of the Nation Outcome Scales (HoNOS, hetero-assessment)
Treatment compliance between groups | 18 months
  item 13 of the Health of the Nation Outcome Scales (HoNOS, hetero-assessment)
Treatment compliance between groups | 2 years
  item 13 of the Health of the Nation Outcome Scales (HoNOS, hetero-assessment)
Treatment compliance between groups | 2.5 years
  item 13 of the Health of the Nation Outcome Scales (HoNOS, hetero-assessment)
Treatment compliance between groups | 3 years
  item 13 of the Health of the Nation Outcome Scales (HoNOS, hetero-assessment)
Adherence to treatment | 1 year
  Medication Adherence Rating Scale (MARS, self-administered questionnaire)
Adherence to treatment | 2 years
  Medication Adherence Rating Scale (MARS, self-administered questionnaire)
Adherence to treatment | 3 years
  Medication Adherence Rating Scale (MARS, self-administered questionnaire)
Therapeutic alliance | 1 year
  Working Alliance Inventory-Short Revised (WAI-SR, self-administered questionnaire)
Therapeutic alliance | 2 years
  Working Alliance Inventory-Short Revised (WAI-SR, self-administered questionnaire)
Therapeutic alliance | 3 years
  Working Alliance Inventory-Short Revised (WAI-SR, self-administered questionnaire)
Patient awareness of disorders and of the need for treatment | 1 year
  Birchwood Insight Scale (BIS, self-administered questionnaire)
Patient awareness of disorders and of the need for treatment | 2 years
  Birchwood Insight Scale (BIS, self-administered questionnaire)
Patient awareness of disorders and of the need for treatment | 3 years
  Birchwood Insight Scale (BIS, self-administered questionnaire)
Assessment of addictive comorbidities | Inclusion
  semi-structured clinical interview for DSM (SCID)
Assessment of addictive comorbidities | 3 years
  semi-structured clinical interview for DSM (SCID)
Assessment of tobacco, alcohol and drug use | Every 6 months from inclusion
  Alcohol, Smoking and Substance Involvement Screening Test (ASSIST)
Evaluation of the clinical impact of the intervention between groups | Every 6 months from inclusion
  Clinical Global Impression questionnaire (CGI)
Psychotic and general symptoms | Every 6 months from inclusion
  Positive and Negative Symptom Scale (PANSS)
Depressive symptoms | Every 6 months from inclusion
  Calgary Depression Scale for Schizophrenia (CDSS)
Self- and hetero-aggressive behaviors | Every 6 months from inclusion
  according to Health of the Nation Outcome Scales (HoNOS) items 1 and 2
Reported adverse events | Inclusion
  death by suicide, attempted suicide or self-injurious acts, hetero-aggressive acts according to the medical record and investigated if score greater than or equal to 3 on items 1 and 2 of the HoNOS
Reported adverse events | 6 months
  death by suicide, attempted suicide or self-injurious acts, hetero-aggressive acts according to the medical record and investigated if score greater than or equal to 3 on items 1 and 2 of the HoNOS
Reported adverse events | 1 year
  death by suicide, attempted suicide or self-injurious acts, hetero-aggressive acts according to the medical record and investigated if score greater than or equal to 3 on items 1 and 2 of the HoNOS
Reported adverse events | 18 months
  death by suicide, attempted suicide or self-injurious acts, hetero-aggressive acts according to the medical record and investigated if score greater than or equal to 3 on items 1 and 2 of the HoNOS
Reported adverse events | 2 years
  death by suicide, attempted suicide or self-injurious acts, hetero-aggressive acts according to the medical record and investigated if score greater than or equal to 3 on items 1 and 2 of the HoNOS
Reported adverse events | 2.5 years
  death by suicide, attempted suicide or self-injurious acts, hetero-aggressive acts according to the medical record and investigated if score greater than or equal to 3 on items 1 and 2 of the HoNOS
Reported adverse events | 3 years
  death by suicide, attempted suicide or self-injurious acts, hetero-aggressive acts according to the medical record and investigated if score greater than or equal to 3 on items 1 and 2 of the HoNOS
Current suicidal ideations | Inclusion
  Calgary Depression Scale for Schizophrenia (CDSS)
Current suicidal ideations | 6 months
  Calgary Depression Scale for Schizophrenia (CDSS)
Current suicidal ideations | 1 year
  Calgary Depression Scale for Schizophrenia (CDSS)
Current suicidal ideations | 18 months
  Calgary Depression Scale for Schizophrenia (CDSS)
Current suicidal ideations | 2 years
  Calgary Depression Scale for Schizophrenia (CDSS)
Current suicidal ideations | 2.5 years
  Calgary Depression Scale for Schizophrenia (CDSS)
Current suicidal ideations | 3 years
  Calgary Depression Scale for Schizophrenia (CDSS)
Assess the impact of the intervention on socio-professional functioning and quality of life | Inclusion
  Socio-demographic data updated every 6 months: living conditions (housing, entourage, income), level of education and/or professional situation
Assess the impact of the intervention on socio-professional functioning and quality of life | 6 months
  Socio-demographic data updated every 6 months: living conditions (housing, entourage, income), level of education and/or professional situation
Assess the impact of the intervention on socio-professional functioning and quality of life | 1 year
  Socio-demographic data updated every 6 months: living conditions (housing, entourage, income), level of education and/or professional situation
Assess the impact of the intervention on socio-professional functioning and quality of life | 18 months
  Socio-demographic data updated every 6 months: living conditions (housing, entourage, income), level of education and/or professional situation
Assess the impact of the intervention on socio-professional functioning and quality of life | 2 years
  Socio-demographic data updated every 6 months: living conditions (housing, entourage, income), level of education and/or professional situation
Assess the impact of the intervention on socio-professional functioning and quality of life | 2.5 years
  Socio-demographic data updated every 6 months: living conditions (housing, entourage, income), level of education and/or professional situation
Assess the impact of the intervention on socio-professional functioning and quality of life | 3 years
  Socio-demographic data updated every 6 months: living conditions (housing, entourage, income), level of education and/or professional situation
Social and occupational functioning | Inclusion
  Social and Occupational Functioning Assessment Scale (SOFAS)
Social and occupational functioning | 6 months
  Social and Occupational Functioning Assessment Scale (SOFAS)
Social and occupational functioning | 1 year
  Social and Occupational Functioning Assessment Scale (SOFAS)
Social and occupational functioning | 18 months
  Social and Occupational Functioning Assessment Scale (SOFAS)
Social and occupational functioning | 2 years
  Social and Occupational Functioning Assessment Scale (SOFAS)
Social and occupational functioning | 2.5 years
  Social and Occupational Functioning Assessment Scale (SOFAS)
Social and occupational functioning | 3 years
  Social and Occupational Functioning Assessment Scale (SOFAS)
Social functioning | Inclusion
  Health of the Nation Outcome Scales
Social functioning | 6 months
  Health of the Nation Outcome Scales
Social functioning | 1 year
  Health of the Nation Outcome Scales
Social functioning | 18 months
  Health of the Nation Outcome Scales
Social functioning | 2 years
  Health of the Nation Outcome Scales
Social functioning | 2.5 years
  Health of the Nation Outcome Scales
Social functioning | 3 years
  Health of the Nation Outcome Scales
Psychosocial functioning | Inclusion
  Quality of Life Scale (QLS) - semi-structured interview
Psychosocial functioning | 6 months
  Quality of Life Scale (QLS) - semi-structured interview
Psychosocial functioning | 1 year
  Quality of Life Scale (QLS) - semi-structured interview
Psychosocial functioning | 18 months
  Quality of Life Scale (QLS) - semi-structured interview
Psychosocial functioning | 2 years
  Quality of Life Scale (QLS) - semi-structured interview
Psychosocial functioning | 2.5 years
  Quality of Life Scale (QLS) - semi-structured interview
Psychosocial functioning | 3 years
  Quality of Life Scale (QLS) - semi-structured interview
Functioning | Inclusion
  Schizophrenia Quality of Life Scale Revision 4: self-administered questionnaire
Functioning | 6 months
  Schizophrenia Quality of Life Scale Revision 4: self-administered questionnaire
Functioning | 1 year
  Schizophrenia Quality of Life Scale Revision 4: self-administered questionnaire
Functioning | 18 months
  Schizophrenia Quality of Life Scale Revision 4: self-administered questionnaire
Functioning | 2 years
  Schizophrenia Quality of Life Scale Revision 4: self-administered questionnaire
Functioning | 2.5 years
  Schizophrenia Quality of Life Scale Revision 4: self-administered questionnaire
Functioning | 3 years
  Schizophrenia Quality of Life Scale Revision 4: self-administered questionnaire
Quality of life of users (patient and family) | 1 year
  World Health Organization Quality of Life brief (WHOQOL-brief)
Quality of life of users (patient and family) | 2 years
  World Health Organization Quality of Life brief (WHOQOL-brief)
Quality of life of users (patient and family) | 3 years
  World Health Organization Quality of Life brief (WHOQOL-brief)
Health-related quality of life | 1 year
  EuroQol-5D 3 level version (EQ-5D-35L)
Health-related quality of life | 2 years
  EuroQol-5D 3 level version (EQ-5D-35L)
Health-related quality of life | 3 years
  EuroQol-5D 3 level version (EQ-5D-35L)
Quality of life of relatives | 1 year
  caregiver schizophrenia quality of life questionnaire (S-CGQoL)
Quality of life of relatives | 2 years
  caregiver schizophrenia quality of life questionnaire (S-CGQoL)
Quality of life of relatives | 3 years
  caregiver schizophrenia quality of life questionnaire (S-CGQoL)
Cost-outcome type ratio | 3 years
  the ratio of the difference in costs between the two strategies divided by the difference in QALYs. This ratio measures the cost per life-year gained in full health, i.e. a cost per QALY. This indicator is obtained by weighting the time spent in each health state h by the utility of that health state measured by the EQ-5D
Cost of care | 3 years
  assessed from a community perspective (health care system, out-of-pocket expenses, caregivers)
Budget impact analysis between strategies | 3 years
  National estimates of avoided costs, care consumption and the cost of implementing the system in the two management strategies
Psychiatric assessment | Inclusion
  Structured Clinical Interview for DSM
Psychiatric assessment | 3 years
  Structured Clinical Interview for DSM
Patient age | Inclusion
Patient sex | Inclusion
Current patient professional/training situation | Over the study until 3 years
  working or studying
Financial situation | Over the study until 3 years
Care pathways taken by patient | Over the study until 3 years
  specialist care sought
Duration of non-treated psychosis | Inclusion
  Interval between start of psychotic symptoms and start of sufficient antipsychotic treatment
Personal and family psychiatric history | Inclusion
Social and academic function | Inclusion
  Premorbid Adjustment Scale
Medical treatment received | Until 3 years
Cerebral imagery | Inclusion
  Normal/abnormal
Cerebral imagery | 1 year
  Normal/abnormal
Cerebral imagery | 2 years
  Normal/abnormal
IQ profile | Inclusion
  Homogenous/heterogenous
IQ profile | 1 year
  Homogenous/heterogenous
IQ profile | 2 years
  Homogenous/heterogenous
IQ | Inclusion
  value
IQ | 1 year
  value
IQ | 2 years
  value
BMI | Inclusion
  kg/m2
BMI | 1 year
  kg/m2
BMI | 2 years
  kg/m2
Fasting glycemia | Inclusion
  mmol/l
Fasting glycemia | 1 year
  mmol/l
Fasting glycemia | 2 years
  mmol/l
Lipid assessment | Inclusion
  Normal/abnormal
Lipid assessment | 1 year
  Normal/abnormal
Lipid assessment | 2 years
  Normal/abnormal
Whole blood count | Inclusion
  Normal/abnormal
Whole blood count | 1 year
  Normal/abnormal
Whole blood count | 2 years
  Normal/abnormal
Electrolytes | Inclusion
  Normal/abnormal
Electrolytes | 1 year
  Normal/abnormal
Electrolytes | 2 years
  Normal/abnormal
Neurological exam | Inclusion
  Normal/abnormal
Neurological exam | 1 year
  Normal/abnormal
Neurological exam | 2 years
  Normal/abnormal
Cardiovascular exam | Inclusion
  Normal/abnormal
Cardiovascular exam | 1 year
  Normal/abnormal
Cardiovascular exam | 2 years
  Normal/abnormal
Morphological exam | Inclusion
  Normal/abnormal
Morphological exam | 1 year
  Normal/abnormal
Morphological exam | 2 years
  Normal/abnormal
Hepatic exam | Inclusion
  Normal/abnormal
Hepatic exam | 1 year
  Normal/abnormal
Hepatic exam | 2 years
  Normal/abnormal
Presence of neurometabolic disease | Inclusion
  Yes/no
Presence of neurometabolic disease | 1 year
  Yes/no
Presence of neurometabolic disease | 2 years
  Yes/no
Electrocardiogram | Inclusion
  Normal/abnormal
Electrocardiogram | 1 year
  Normal/abnormal
Electrocardiogram | 2 years
  Normal/abnormal
C-reactive protein | Inclusion
  mg/l
C-reactive protein | 1 year
  mg/l
C-reactive protein | 2 years
  mg/l
thyroid-stimulating hormone | Inclusion
  mUI/l
thyroid-stimulating hormone | 1 year
  mUI/l
thyroid-stimulating hormone | 2 years
  mUI/l
Cortisol | Inclusion
  nmol/l
Cortisol | 1 year
  nmol/l
Cortisol | 2 years
  nmol/l
Adverse events | Inclusion
  Any of the following (yes/no): Neurological symptoms, overweight, metabolic syndrome, sexual dysfunction, fatigue, salivation dysfunction, other
Adverse events | 1 year
  Any of the following (yes/no): Neurological symptoms, overweight, metabolic syndrome, sexual dysfunction, fatigue, salivation dysfunction, other
Adverse events | 2 years
  Any of the following (yes/no): Neurological symptoms, overweight, metabolic syndrome, sexual dysfunction, fatigue, salivation dysfunction, other
Non-medical treatment received | Until 3 years
  Psychosocial/psychotherapy interventions
In the experimental group: case management according to good practice guidelines | End of follow-up (3 years)
  EPPIC Model Integrity Tool (80 items with subscores)
In the experimental group: Conformity of case management | End of study (5 years)
  Index of Fidelity to Assertive Community Treatment (16 criteria of conformity for three dimensions)
In the experimental group: conformity to TIDieR checklist in each patient | Month 3
  TIDieR checklist-patient
In the experimental group: conformity to TIDieR checklist in each patient | Month 6
  TIDieR checklist-patient
In the experimental group: conformity to TIDieR checklist in each patient | 1 year
  TIDieR checklist-patient
In the experimental group: conformity to TIDieR checklist in each patient | 18 Months
  TIDieR checklist-patient
In the experimental group: conformity to TIDieR checklist in each patient | 2 years
  TIDieR checklist-patient
In the experimental group: conformity to TIDieR checklist in each patient | 30 Months
  TIDieR checklist-patient
In the experimental group: conformity to TIDieR checklist in each patient | 3 years
  TIDieR checklist-patient
In the experimental group: conformity to TIDieR checklist in each center | Annually until end of study (5 years)
  Customized TIDieR checklist-center
Satisfaction of patients and their families | 1 year
  Client Satisfaction Questionnaire (CSQ)-8
Satisfaction of patients and their families | 2 years
  Client Satisfaction Questionnaire (CSQ)-8
Satisfaction of patients and their families | 3 years
  Client Satisfaction Questionnaire (CSQ)-8
Satisfaction of participants receiving help from a health coordinator | End of follow-up (3 years)
  7-item custom questionnaire with free answer section

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie Schandrin, Principal Investigator — CHU Nimes
Locations (6):
- France (6):
  - CHU de TOULOUSE, Toulouse, Choisir Une Région
  - CH Saint Marie Clermont-Ferrand, Clermont-Ferrand
  - CHU de Montpellier, Montpellier
  - CHU Nice, Nice
  - CHU de Nîmes, Nîmes
  - Centre Hospitalier Léon-Jean Grégory, Thuir

REFERENCES:
- [Background] Schandrin A, Jourdan J, Chkair S, Bouvet S, Fabbro-Peray P, Abbar M; PEPsy-CM working group. PEPsy-CM study protocol: impact of a 3-year program for early psychosis based on case-management on relapse rate, a French multicenter randomized trial. BMC Psychiatry. 2025 May 15;25(1):488. doi: 10.1186/s12888-025-06940-y. PMID 40375175